CLINICAL TRIAL: NCT01148615
Title: A Phase I, Dose Escalation Study of the Safety, Tolerability, and Pharmacokinetics of Intravenous Aflibercept in Combination With Intravenous Docetaxel Administrated Every 3 Weeks in Chinese Patients With Advanced Solid Malignancies
Brief Title: A Study of Intravenous Aflibercept With Docetaxel in Chinese Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCD11382; U1111-1116-5774 (Other: UTN)
Record Dates: First submitted 2010-06-21; First posted 2010-06-22 (Estimated); Last update posted 2012-01-13 (Estimated); Status verified 2012-01

CONDITIONS: Neoplasm Malignant
MeSH Terms: conditions — Neoplasms | interventions — aflibercept; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aflibercept/ docetaxel (Experimental): Patients with advanced cancer will receive different doses of aflibercept in combination with approved dose of docetaxel.
  Aflibercept 4 or 6mg/kg over 1 hour IV immediately followed by Docetaxel 75mg/m2 IV over 1 hour on Day 1, every 3 weeks
  Interventions: Drug: Aflibercept (AVE0005); Drug: Docetaxel (XRP6976)

INTERVENTIONS:
Drug: Aflibercept (AVE0005) — Pharmaceutical form: solution for infusion
  Route of administration: intravenous
Drug: Docetaxel (XRP6976) — Pharmaceutical form: solution for infusion
  Route of administration: intravenous

SUMMARY:
Primary Objective:

* To confirm the dose of aflibercept in western studies by assessing the dose-limiting toxicity (DLT) of intravenous (IV) aflibercept when administered in combination with docetaxel given intravenously every 3 weeks in Chinese patients with solid tumors.

Secondary Objectives:

* To assess the safety profile of intravenous (IV) aflibercept when administered in combination with docetaxel
* To determine the pharmacokinetics of IV aflibercept and docetaxel when administered in combination
* To make a preliminary assessment of antitumor effects of the combination of docetaxel plus aflibercept in patients with evaluable disease
* To evaluate the immunogenicity of IV aflibercept
* To measure endogenous free Vascular Endothelial Growth Factor (VEGF)

DETAILED DESCRIPTION:
The duration of screening, treatment, and follow-up are within 21 days, 3 weeks/cycle, and 90 days after the last aflibercept administration. Patients will be administered aflibercept in combination with docetaxel until when/if a definitive treatment discontinuation criterion is met such as progressive disease, unacceptable toxicity or patient refusal to continue.

ELIGIBILITY:
Inclusion criteria :

* Histologically or cytologically confirmed solid malignancy that metastatic or unresectable for which standard curative measures do not exist, but for which docetaxel treatment is appropriate.

Exclusion criteria :

* Squamous histology/cytology lung cancer
* Need for a major surgical procedure or radiation therapy during the study
* Treatment with chemotherapy, hormonal therapy, radiotherapy, surgery, or an investigational agent within 28 days
* Cumulative radiation therapy to >25% of the total bone marrow
* History of brain metastases
* Eastern Cooperative Oncology Group(ECOG)>1
* Prior docetaxel treatment but have not been appropriate for safety reasons
* Inadequate organ and bone marrow function
* Uncontrolled hypertension
* Evidence of clinically significant bleeding diathesis or underlying coagulopathy

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-07; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) | 3 weeks (cycle 1)

SECONDARY OUTCOMES:
Global safety profile based on treatment emergent adverse events, serious adverse events, and laboratory abnormalities | Up to 30 days after last administration within a maximum follow up of 18 months
Pharmacokinetic parameters of aflibercept | up to last aflibercept administration +90 days
Pharmacokinetic parameters of docetaxel | cycle 1
Tumor response rate as calculated by the Response Evaluation Criteria in Solid Tumors (RECIST v1.1) | up to a maximum follow-up of 18 months
Immunogenicity of Aflibercept | up to last aflibercept administration+90 days
Endogenous free VEGF | up to last aflibercept administration+30 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Investigational Site Number 156001, Guangzhou, China

REFERENCES:
- [Derived] Huang Y, Zou BY, Zhao LP, Zhao HY, Zhao YY, Xue C, Zhang JW, Xu F, Chen LK, Liu JL, Hu ZH, Wu X, Zhang J, Ma YX, Wei CL, Ma Y, Zhang L. Phase I dose-escalation study of aflibercept plus docetaxel in nasopharyngeal carcinoma and other solid tumors. Future Oncol. 2014 Dec;10(16):2579-91. doi: 10.2217/fon.14.206. PMID 25531046